CLINICAL TRIAL: NCT01388179
Title: Deep rTMS(Repetitive Transcranial Magnetic Stimulation) for Treatment of Autism Symptoms in Children With Low Functioning ASD (Autism Spectrum Disorders)
Brief Title: Deep rTMS (Repetitive Transcranial Magnetic Stimulation)for Treatment of Autism Symptoms in Children.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to stop the study
Sponsor: Brainsway (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS-AUTISM
Record Dates: First submitted 2011-06-27; First posted 2011-07-06 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Autism
Keywords: Autism; TMS
MeSH Terms: conditions — Autistic Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real rTMS treatment (Active Comparator): low-frequency rTMS to the left DLPFC (Dorsa-Lateral Pre-Frontal Cortex) prior to high-frequency deep rTMS to the FFA (Fusi-Form Area) through the STS(Superior Temporal Sulcus).
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham rTMS treatment (Sham Comparator): Sham coil which simulate the real coil action
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — low-frequency rTMS to the left DLPFC prior to high-frequency deep rTMS to the FFA through the STS.

SUMMARY:
Autism is a developmental disorder characterized by abnormalities in speech and communication, impaired social functioning, and repetitive behaviors and interests. The term "Autism spectrum disorders" or ASD is often used to include autistic disorder, Asperger syndrome and pervasive developmental disorder-not otherwise specified (PDD-NOS). Epidemiological research suggests that ASDs affect at least 60 per 10,000 youth, with estimates as high as 120 per 10,000.

Severity of autistic features is not easily defined and the use of different diagnostic tools compounds the ability to lay a clear cut definition. It is, though, generally accepted that children with autism and normal IQ (>70) are "high functioning" regardless of the severity of their autistic features. The investigators will use the terms "autism" and "ASD" interchangeably, and the term "low functioning autism" will be used to describe those children with autism who have, or are presumed to have, IQ<70.

The pathophysiology of autism has been studied extensively in the last decade. Abnormal neuronal connectivity has been implicated in a growing body of research. In addition, areas of over and/or under neuronal activation have been detected on functional MRI(Magnetic Resonance Imaging).

Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive technique that allows to affect brain activity. The pulses are administered by passing high currents through an electromagnetic coil placed adjacent to a patient's scalp. The pulses induce an electric field in the underlying brain tissue. When the induced field is above a certain threshold, and is directed in an appropriate orientation relative to the brain's neuronal pathways, localized axonal depolarizations are produced, thus activating the neurons in the relevant brain structure.

rTMS has been studied in individuals with high functioning autism. rTMS treatment was found to have an electrophysiological effect and to reduce repetitive behaviors and improved social functioning.

In the context of existing pilot data suggesting effect of rTMS treatment in individuals with high functioning autism, the investigators propose a pilot study to assess the efficacy of rTMS in children and adolescents with low functioning autism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 10-19 years of age. Although we assume that the effect of rTMS may be greater in younger children, in whom secondary behavioral issues may be less established, the study will focus on children older than age 10 years for 2 reasons:

   i. Some cooperation is needed by the children to undergo a rTMS treatment. ii. We would like to establish the efficacy and safety profile of this treatment in older children with autism before we expose younger children, who may need sedation, to it.
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision criteria. Children will have had a diagnosis of ASD prior to the study given by a pediatric neurologist, child psychiatrist or developmental pediatrician. Diagnosis will be confirmed by Autism Diagnostic Observation Schedule (ADOS-G) and Autism Diagnostic Interview (ADI-R)
3. VABS-II score in the low-very low range. This study is recruiting low functioning individuals with Autism. Although some of the assessment tools (i.e. ASRS) are standardized and validated on individuals without intellectual disabilities, there has been experience using these tools in children with autism in all intellectual levels. In addition, because we are measuring a change over time and not endorsing a diagnosis, we feel that using these tools is sufficient.
4. Have normal physical examination.
5. TAS (Transcranial magnetic stimulation Safety Screen questionnaire) is negative or mitigated as per parent prior to the study.

Exclusion Criteria:

1. Patients born prior to 37 weeks gestational age.
2. Patients with any primary psychiatric diagnosis other than autism at screening.
3. Patients with a medical history of neurological disease, including, but not limited to, movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal MRI/structural lesion of the brain or a history of traumatic brain injury.
4. Patients with a medical history of epilepsy/seizure disorder
5. Patients with a family history of epilepsy in a first degree relative (parent or sibling)
6. Patients with a medical condition other then autism
7. Patients prescribed with psychoactive medication(s) less then 4 weeks prior to joining the study.
8. Patients with a medical history head trauma associated with prolonged loss of consciousness.
9. History of metal foreign body in the head, excluding oral devices
10. History of known anatomical brain abnormality
11. Hearing loss
12. participation in an ongoing other interventional study

Discontinuation criteria:

1. The patient or legal guardian refuses to continue
2. The RC decides that the patient is not suitable to continue the study
3. Severe side effects

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01-23 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
CGI-I(clinical global impression-I) as a measure for social functioning | 90 days from first day of treatment
  rTMS treatment will be superior to sham treatment in improving social functioning (using the CGI-I Social) in children and adolescents with ASD.
ASRS (Adult ADHD Self Report Scale) as a measure for social awareness and social motivation | 90 days from first day of treatment
  rTMS treatment will be superior to sham treatment in improving social awareness and social motivation (using the ASRS) in children and adolescents with ASD.
Facial recognition test as a measure for preference to faces vs. objects | 90 days from first day of treatment
  rTMS treatment will be superior to sham treatment in increasing preference to faces vs. objects as measured by a facial recognition test, in children and adolescents with ASD.

SECONDARY OUTCOMES:
PLS-4(Preschool Language Scale - 4 ) as a measure for language impairment. | 90 days from first treatment
  rTMS treatment will be superior to sham treatment in the treatment of language impairment (using the PLS-4 Hebrew language assessment)
BASC (Behavior Assessment System for Children) as a measure for anxiety | 90 days from first day of treatment
  rTMS will be superior to sham in the treatment of the associated autism symptom domains of anxiety (BASC-anxiety subscale)
ABC (Autism Behavior Checklist)as a measure for repetitive behaviors | 90 days from first day of treatment
  rTMS treatment will be superior to sham treatment in the treatment of repetitive behaviors (using the Aberrant Behavior Checklist -ABC) in children and adolescents with ASD.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel